CLINICAL TRIAL: NCT02323971
Title: Impact of Renal Function on Ticagrelor-Induced Antiplatelet Effects in Coronary Artery Disease Patients
Acronym: Ticagrelor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: FFI-TIC-2014-01
Record Dates: First submitted 2014-12-12; First posted 2014-12-24 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ticagrelor

SUMMARY:
Dual antiplatelet therapy consisting in aspirin and clopidogrel is the cornerstone of the treatment of the prevention of the thrombotic events in patients with coronary artery disease (CAD), showing a reduction in adverse events.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting in aspirin and clopidogrel is the cornerstone of the treatment of the prevention of the thrombotic events in patients with coronary artery disease (CAD), showing a reduction in adverse events . However, there is a considerable number of patients who continue to have recurrent ischemic events despite this regimen . In fact, in the last years several clinical factors have been associated with impaired clopidogrel-induced effects. Moreover, these clinical factors are strongly related with the presence of high on-treatment platelet reactivity (HPR), which is also associated with the occurrence of adverse thrombotic events, including stent thrombosis, despite correct treatment compliance. Diabetes mellitus, acute coronary syndromes, obesity or chronic kidney disease (CKD) are common examples . This observation encourages the search for new more potent antiplatelet therapies. A new P2Y12 receptor antagonist, ticagrelor, has been approved for clinical use . Ticagrelor is a new non-thienopyridine, a cyclopentyltriazolo-pyrimidine (CPTP), direct acting reversible P2Y12 antagonist. This compound has a more favorable pharmacokinetic (PK) and pharmacodynamics (PD) profile than clopidogrel , which has translated into better clinical outcomes in patients with acute coronary syndrome (ACS) in a recent large, international clinical trial . Interestingly, ticagrelor has showed an impressive clinical benefit in patients with CKD in comparison with those patients without renal impairment .

CKD is highly associated with an increased risk of atherothrombotic events, including stent thrombosis, in patients with CAD . PD studies have shown that patients with impaired renal function are characterized by reduced clopidogrel-induced antiplatelet effects and higher rates of HPR compared with patients with preserved renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with moderate-high risk non-STEACS defined according the current guidelines
* Patients received a loading dose or under chronic treatment with aspirin (100 mg per day) as per standard of care
* Age between 18 and 80 years old
* BMI between 18 and 35 kg/m2
* Provide written informed consent prior to any study specific procedures

Exclusion Criteria:

* History of hemorrhagic stroke or intracranial bleeding
* Known allergies to aspirin, ticagrelor, or clopidogrel
* On treatment with oral anticoagulation (Coumarin derivate, dabigatran, rivaroxaban, apixaban)
* Hemoglobin <10 gm/dL
* Platelet count <80x106/mL
* Blood dyscrasias, active bleeding or hemodynamic instability.
* Patients on hemodialysis or peritoneal dialysis, a change in estimated glomerular filtration rate (eGFR) greater than 15 mL/min within 90 days prior to enrollment, or estimated glomerular filtration rate (eGFR) lower than 15 mL/min/1.73m2
* Patients with known infectious diseases or neoplasia
* Baseline ALT >2.5 times the upper limit of normal
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection
* Drugs interfering with 2C19 metabolism (to avoid interaction with clopidogrel): fluconazole (Diflucan), ketoconazole (Nizoral), voriconazole (VFEND), etravirine (Intelence), felbamate (Felbatol), fluoxetine (Prozac, Serafem, Symbyax), fluvoxamine (Luvox), and ticlopidine (Ticlid). Since omeprazole is the most used proton-pump inhibitor in our clinical environment, we will keep the same prescription rate in both groups to avoid differences results from this described interaction
* Drugs interfering CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin
* Pregnant females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD and with normal renal function
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
platelet reactivity units | 7+2 days of treatment
  The primary endpoint is the comparison of the platelet reactivity units (PRU) values determined by VerfifyNow-P2Y12 system between normal renal function and CKD patients after 7±2 days of concomitant treatment with ticagrelor.

SECONDARY OUTCOMES:
platelet reactivity profiles after loading dose of ticagrelor | 30 min, 1, 2, 4 and 6 hours
  To evaluate platelet reactivity profiles after loading dose of ticagrelor using a 180 mg loading dose at 30 min, 1, 2, 4 and 6 hours, and comparing CKD to non-CKD patients as measured with VerifyNow-P2Y12 system.
platelet reactivity profiles after 180 mg loading dose to ticagrelor usin MEA | 30 min, 1, 2, 4 and 6 hours
  To analyze platelet reactivity profiles after 180 mg loading dose to ticagrelor using MEA, at 30 min, 1, 2, 4 and 6 hours and after 90 mg b.i.d maintenance dose of ticagrelor at 7±2 days.
ticagrelor active metabolite levels | 30 min, 1, 2, 4 and 6 hours
  To assess ticagrelor active metabolite levels after loading dose of ticagrelor using a 180 mg loading dose at 30 min, 1, 2, 4 and 6 hours, and comparing CKD to non-CKD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tello-Montoliu MD Antonio, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, Murcia, Spain